CLINICAL TRIAL: NCT06029920
Title: The Effect of Overground Walking on the Increase of Brain-Derived Neurotrophic Factor Levels, IL-6, HS-CRP, Cognitive Function, and Quality of Life in the Elderly
Brief Title: Influence of Overground Walking on Biomarkers, Cognitive Function, and Quality of Life in Elderly With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Irma Ruslina Defi, Principal Investigator, Universitas Padjadjaran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IKFR.2023.08.01
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cognitive Impairment; Aging
Keywords: Exercise; Rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects (Experimental)
  Interventions: Other: Overground Walking

INTERVENTIONS:
Other: Overground Walking — Walk on a flat surface for a distance of 15 meters, with a duration of 20 minutes, increasing by 5 minutes each week until the target heart rate is achieved during the exercise, for 8 weeks.

SUMMARY:
The purpose of this research is to investigate the impact of overground walking as a part of a rehabilitation program on the increase in Brain-derived neurotrophic factor (BDNF) levels, decrease in IL-6 levels, decrease in hs-CRP levels, improvement in cognitive function, and enhancement of quality of life (QOL) in older people with mild cognitive impairment. These findings are anticipated to contribute to the efforts to elevate BDNF levels, cognitive function, and QOL while reducing IL-6 and hsCRP levels in the elderly with mild cognitive impairment.

DETAILED DESCRIPTION:
This research employs a quasi-experimental research design using a Pretest-Posttest Design approach. The Pretest-Posttest method is executed by assessing before and after the intervention within the same group.

All research subjects receive the same treatment, which involves participating in an overground walking program on a flat surface. The selected research subjects are provided with an explanation of the research's objectives and benefits and the exercise and examination procedures, then sign the informed consent.

Research subjects are instructed to walk on a flat surface for a distance of 15 meters, with a duration of 20 minutes, increasing by 5 minutes each week until the target heart rate is achieved during the exercise. After an 8-week post-intervention period, research subjects will undergo a follow-up examination.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment (MoCA INA Score 19-25 out of 30
* Barthel Index Score 20
* Geriatric Depression Scale Score ≤ 5
* Timed Up and Go Test < 15 seconds)
* Capable of comprehending verbal and written instructions
* Capable of walking unassisted

Exclusion Criteria:

* The presence of hearing impairment that could hinder the subject from receiving verbal instructions,
* The presence of uncorrected visual impairment
* Having musculoskeletal disorders
* Receiving other rehabilitation programs,
* Presence of diseases causing cognitive impairment
* Severe joint diseases such as osteoarthritis and rheumatoid arthritis that may worsen during exercise or could pose difficulties in carrying out the exercise program,
* Severe cardiovascular diseases as diagnosed by a Cardiologist

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
BDNF | 8 weeks
  Brain-derived neurotrophic factor level
IL6 | 8 weeks
  Interleukin-6 level
hsCRP | 8 weeks
  hs-CRP level
MoCAINA | 8 weeks
  MONTREAL COGNITIVE ASSESSMENT INDONESIA
ADQOL | 8 weeks
  Alzheimer disease Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing Home, Bandung, West Java, Indonesia

REFERENCES:
- [Background] Amieva H, Letenneur L, Dartigues JF, Rouch-Leroyer I, Sourgen C, D'Alchee-Biree F, Dib M, Barberger-Gateau P, Orgogozo JM, Fabrigoule C. Annual rate and predictors of conversion to dementia in subjects presenting mild cognitive impairment criteria defined according to a population-based study. Dement Geriatr Cogn Disord. 2004;18(1):87-93. doi: 10.1159/000077815. Epub 2004 Apr 14. PMID 15087583
- [Background] Barrios H, Narciso S, Guerreiro M, Maroco J, Logsdon R, de Mendonca A. Quality of life in patients with mild cognitive impairment. Aging Ment Health. 2013;17(3):287-92. doi: 10.1080/13607863.2012.747083. Epub 2012 Dec 7. PMID 23215827
- [Background] Bavelier D, Neville HJ. Cross-modal plasticity: where and how? Nat Rev Neurosci. 2002 Jun;3(6):443-52. doi: 10.1038/nrn848. PMID 12042879
- [Background] Burkhalter TM, Hillman CH. A narrative review of physical activity, nutrition, and obesity to cognition and scholastic performance across the human lifespan. Adv Nutr. 2011 Mar;2(2):201S-6S. doi: 10.3945/an.111.000331. Epub 2011 Mar 10. PMID 22332052
- [Background] Chieffi S, Messina G, Villano I, Messina A, Valenzano A, Moscatelli F, Salerno M, Sullo A, Avola R, Monda V, Cibelli G, Monda M. Neuroprotective Effects of Physical Activity: Evidence from Human and Animal Studies. Front Neurol. 2017 May 22;8:188. doi: 10.3389/fneur.2017.00188. eCollection 2017. PMID 28588546
- [Background] Dik M, Deeg DJ, Visser M, Jonker C. Early life physical activity and cognition at old age. J Clin Exp Neuropsychol. 2003 Aug;25(5):643-53. doi: 10.1076/jcen.25.5.643.14583. PMID 12815502
- [Background] Espino DV, Lichtenstein MJ, Palmer RF, Hazuda HP. Ethnic differences in mini-mental state examination (MMSE) scores: where you live makes a difference. J Am Geriatr Soc. 2001 May;49(5):538-48. doi: 10.1046/j.1532-5415.2001.49111.x. PMID 11380745
- [Background] Harada CN, Natelson Love MC, Triebel KL. Normal cognitive aging. Clin Geriatr Med. 2013 Nov;29(4):737-52. doi: 10.1016/j.cger.2013.07.002. PMID 24094294
- [Background] Shams A, Nobari H, Afonso J, Abbasi H, Mainer-Pardos E, Perez-Gomez J, Bayati M, Bahrami A, Carneiro L. Effect of Aerobic-Based Exercise on Psychological Well-Being and Quality of Life Among Older People: A Middle East Study. Front Public Health. 2021 Dec 6;9:764044. doi: 10.3389/fpubh.2021.764044. eCollection 2021. PMID 34938705
- [Background] Xue J, Li J, Liang J, Chen S. The Prevalence of Mild Cognitive Impairment in China: A Systematic Review. Aging Dis. 2018 Aug 1;9(4):706-715. doi: 10.14336/AD.2017.0928. eCollection 2018 Aug. PMID 30090658